CLINICAL TRIAL: NCT00130988
Title: Efficacy of a Biopsychosocial Treatment for Somatizing Patients Carried Out by the General Practitioner
Brief Title: DEPENAS: A Psychosocial Intervention for Patients With Medically Unexplained Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Jose María Aiarzaguena, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00/00854
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Somatoform Disorders
Keywords: Somatoform Disorders; Medically unexplained symptoms; Physician-Patient Relations; Primary Health Care; Family Physician; psychosocial therapy; re-attribution of symptoms; cluster randomised controlled trial
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: DEPENAS cognitive and behavioural techniques

SUMMARY:
General practitioners play a key role in the management of one of the most complex problems facing the health care system: the large group of patients with unexplained medical symptoms, but effective treatment strategies are lacking in primary care. The purpose of this study is to compare a new intervention delivered by the general practitioner versus re-attribution of symptoms, which is the currently recommended best treatment for patients with high levels of medically unexplained physical symptoms.

DETAILED DESCRIPTION:
Patients with unexplained medical symptoms are frequently referred to multiple specialists, including psychiatrists, which often prove ineffective. General practitioners play a key role in the management of these patients and techniques of re-attribution of symptoms have been proposed for general practice, but they have only shown partial results in patients with somatised mental disorders who do not believe that their symptoms have a completely physical cause.

Based on the analysis of psychosocial interventions carried out in general practice over the last 10 years by the principal investigator (JMA), the investigators have empirically structured a new sort of intervention, called DEPENAS. This new intervention integrates different psychotherapeutic models. It starts with the attribution of symptoms to a hormonal imbalance (biological aspect) providing a tangible and exculpatory explanation of the patients' symptoms and follows with normalization/justification of any thought/behavior as a logical consequence derived from the personal and family cycle (systemic model). It ends with a proposal for change: to adapt these thoughts, many of them infantile, to objectives of adulthood (transactional model) using cognitive and behavioral techniques in patients ready for change, or paradoxical techniques for non-prepared subjects.

The OBJECTIVE of this randomized clinical trial was to assess the efficacy of this new intervention carried out by family physicians on patients' self-perceived health related quality of life (SF-36). Each doctor randomly allocated to the new intervention group performed six 30-min programmed and standardized sessions with four patients who presented multiple chronic physical symptoms that remained medically unexplained. Health related quality of life was measured at baseline (1 month before starting therapy), after 3 months of the first appointment (once both study groups had completed five sessions), after 8 months (once the intervention was finished) and at 12 months after enrollment.

They will be COMPARED to patients of family doctors randomly assigned to the control group. These doctors also performed six 30-min programmed and standardized sessions, using in this case "re-attribution techniques": reception and explicit acceptance of the patient's symptoms, examination of emotional and psychosocial problems and establishment of a link of the symptoms with identified emotional problems. Patients' outcomes observed in both groups will be compared on an intention to treat basis, and random-effects longitudinal models will be used to estimate the effect of the intervention on quality of life evolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age, who had presented (over the course of their lives) six or more medically unexplained somatic symptoms for female subjects and four or more for male subjects
* At least one of the symptoms would have continued to be present during the last year

Exclusion Criteria:

* Dementia
* Psychotic disorders
* Drug dependence
* Bipolar disorder
* Eating disorders
* Malingering patients
* Patients engaged in psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156
Dates: Start 2001-01; Primary Completion 2002-02 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Aiarzaguena, Dr., Principal Investigator — Basque Health Service

REFERENCES:
- [Background] Aiarzaguena JM, Grandes G, Alonso-Arbiol I, del Campo Chavala JL, Oleaga Fernandez MB, Marco De Juana J. [Bio-psychosocial treatment approach to somatizing patients in primary care: a pilot study]. Aten Primaria. 2002 May 31;29(9):558-61. doi: 10.1016/s0212-6567(02)70637-9. Spanish. PMID 12061987
- [Background] Rosendal M, Olesen F, Fink P. Management of medically unexplained symptoms. BMJ. 2005 Jan 1;330(7481):4-5. doi: 10.1136/bmj.330.7481.4. No abstract available. PMID 15626783
- [Background] Mayou R, Farmer A. ABC of psychological medicine: Functional somatic symptoms and syndromes. BMJ. 2002 Aug 3;325(7358):265-8. doi: 10.1136/bmj.325.7358.265. No abstract available. PMID 12153926
- [Background] Raine R, Haines A, Sensky T, Hutchings A, Larkin K, Black N. Systematic review of mental health interventions for patients with common somatic symptoms: can research evidence from secondary care be extrapolated to primary care? BMJ. 2002 Nov 9;325(7372):1082. doi: 10.1136/bmj.325.7372.1082. PMID 12424170
- [Background] Wileman L, May C, Chew-Graham CA. Medically unexplained symptoms and the problem of power in the primary care consultation: a qualitative study. Fam Pract. 2002 Apr;19(2):178-82. doi: 10.1093/fampra/19.2.178. PMID 11906984
- [Background] Barsky AJ, Borus JF. Somatization and medicalization in the era of managed care. JAMA. 1995 Dec 27;274(24):1931-4. PMID 8568987
- [Background] Aiarzaguena JM, Grandes G, Gaminde I, Salazar A, Sanchez A, Arino J. A randomized controlled clinical trial of a psychosocial and communication intervention carried out by GPs for patients with medically unexplained symptoms. Psychol Med. 2007 Feb;37(2):283-94. doi: 10.1017/S0033291706009536. Epub 2006 Dec 13. PMID 17164029
- [Derived] Aiarzaguena JM, Gaminde I, Grandes G, Salazar A, Alonso I, Sanchez A. Somatisation in primary care: experiences of primary care physicians involved in a training program and in a randomised controlled trial. BMC Fam Pract. 2009 Nov 25;10:73. doi: 10.1186/1471-2296-10-73. PMID 19930729